CLINICAL TRIAL: NCT05812001
Title: The Efficacy of Exergames-acceptance and Commitment Therapy Program for Treatment of Major Depressive Disorder: Comparison With Acceptance and Commitment Therapy Alone and Treatment-as-usual in a Randomized Controlled Trial
Brief Title: Exergames-acceptance and Commitment Therapy Program for Treatment of Major Depressive Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Principal Investigator, Mohammad Farris Iman Leong Bin Abdullah, Medical lecturer, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1679299088
Record Dates: First submitted 2023-03-20; First posted 2023-04-13 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial (RCT) is multicentre, three-armed, parallel-group, double-blind RCT.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be kept unaware of the study's randomization into the designated groups, conducted by a research assistant who is not otherwise involved in the study and concealed in an opaque, sequentially numbered envelope. Therefore, participants will not know which group they are allocated to. In addition, the intervention groups (e-ACT or ACT) and the treatment-as-usual control group will receive equal amount of attention and time from the professional figure who administer the program. The researchers will also be "blinded" for the study since the participants' randomized assignment into the designated groups will be conducted by a research assistant who is not otherwise involved in the study. This project's data collection and analysis will also be conducted by that research assistant who is not otherwise involved in the study or data analysis and who is unaware of the study's hypotheses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exergames-acceptance and commitment therapy (e-ACT) group (Experimental): Exergame is playing of video games that require rigorous physical exercise and are intended as a work-out, such as those in which players race a virtual bicycle on-screen by pedalling a simulator resembling an exercise bike. It not only improve motivation, physical fitness and cognitive function, but it also induces antidepressant effect similar to physical exercise. Acceptance and commitment therapy (ACT) is a third-generation cognitive behavioral approach which uses acceptance and mindfulness processes, and commitment and behavior change processes to produce psychological flexibility. ACT was designed to increase adaptive coping through acceptance, cognitive defusion, mindfulness, and perspective-taking exercises while supporting depression patients in aligning behavior with their personal values. Hence, the combination of both exergame and ACT may provide additional benefit for treatment of depression patients beyond the degree of effectiveness of ACT alone.
  Interventions: Behavioral: Exergames-acceptance and commitment therapy (e-ACT)
- Acceptance and commitment therapy (ACT) group (Active Comparator): It is a third-generation cognitive behavioral approach which uses acceptance and mindfulness processes, and commitment and behavior change processes to produce psychological flexibility. Unlike CBT, which aims to change unhelpful thoughts and feelings, ACT was designed to increase adaptive coping through acceptance, cognitive defusion, mindfulness, and perspective-taking exercises while supporting depression patients in aligning behavior with their personal values. Hence, ACT consists of 8 sessions, one session per week to facilitate depression patients to development and maintenance of health behavioral improvements by targeting internal barriers, such as emotional discomfort and self-defeating thoughts, and by fostering connection and commitment to personal values associated with self-management of positive health behaviors.
  Interventions: Behavioral: Acceptance and commitment therapy (ACT)
- Treatment-as-usual control (TAU) group (No Intervention): The participants in the control group will receive treatment-as-usual in which non-specific ingredients of the psychotherapeutic approach will be administered, such as psychological understanding to the management of an individual patient, identifying current problems, providing opportunities for disclosure, reassurance, and deep breathing exercise. They will be given equal amount of time and attention from the professional figure compared to the intervention groups, whereby they will also attach to an 8-session program (with one session per week for 8 weeks). Each weekly TAU session will be held at the same time (± 2 hours) and at the same venue (in the psychology lab).

INTERVENTIONS:
Behavioral: Exergames-acceptance and commitment therapy (e-ACT) — In the e-ACT training program, participants will perform a 30-minute per session Nintendo-program on TV for three days per week and a 50-minute ACT session per week for 8 weeks which will take place in the psychology labs of AMDI, USM. The ACT session will be held after 30 minutes break following the completion of the final exergame session of the week. Hence, the total duration of each weekly e-ACT training session will be approximately 2 hours. In addition, each weekly e-ACT training session will be held at the same time (± 2 hours) and at the same venue.
  Arms: Exergames-acceptance and commitment therapy (e-ACT) group
Behavioral: Acceptance and commitment therapy (ACT) — As for the ACT intervention, each ACT session will run for 50 minutes, one session per week for 8 weeks. Each weekly ACT session will be held at the same time (± 2 hours) and at the same venue (in the psychology lab).
  Arms: Acceptance and commitment therapy (ACT) group

SUMMARY:
Background: The prevalence of depressive disorder, particularly major depressive disorder is on the rise globally and the use of antidepressant medication for treatment does not usually resulting in full remission. However, combination of antidepressant medication and psychotherapy for treatment of major depressive disorder (MDD) increase the rate of full remission compared to antidepressant monotherapy. This three-armed, parallel-group, double-blind, randomized control trial (RCT) aims to assess and compare the effects of combination of exergame and acceptance and commitment (e-ACT) training programme and ACT only on psychiatric symptoms (depression and anxiety), experiential avoidance (EA), quality of life (QoL), and biomarkers of depression (such as BDNF, CRP, and VEGF) among MDD patients.

Methods: This RCT will recruit 120 patients diagnosed with MDD who will be randomized using stratified permuted block randomization into three groups, which are combined e-ACT training programme, ACT only and treatment-as-usual control groups in a 1:1:1 allocation ratio. The participants in the e-ACT and ACT only intervention groups will undergo once a week intervention sessions for 8 weeks. Assessments will be carried out through three time points, such as the first assessment before intervention began (t0), second assessment immediately after completion of intervention at 8 weeks (t1) and third assessment 24 weeks after completion of intervention (t2). During each assessment, the primary outcome assessed is the severity of depression symptoms, while the secondary outcomes assessed are severity of anxiety symptoms, QoL, EA, and biomarkers of depression.

DETAILED DESCRIPTION:
Objective

General:

To evaluate the efficacy of of exergames-acceptance and commitment therapy (e-ACT) training program compared to acceptance and commitment therapy (ACT) alone or a treatment-as-usual control group.

Specific:

Primary objectives:

(1)To evaluate the efficacy of exergames-acceptance and commitment therapy (e-ACT) training program on reducing severity of depressive symptoms among patients with major depressive disorder compared to ACT only and a control group (treatment-as-usual) across three timelines, such as pre-intervention, immediately post-intervention (8 weeks) and 24 weeks post-intervention.

Secondary objectives:

1. To evaluate the efficacy of exergames-acceptance and commitment therapy (e-ACT) training program on increasing quality of life (QoL) among patients with major depressive disorder compared to ACT only and a control group (treatment-as-usual) across three timelines, such as pre-intervention, immediately post-intervention (8 weeks) and 24 weeks post-intervention.
2. To evaluate the efficacy of exergames-acceptance and commitment therapy (e-ACT) training program on reducing experiential avoidance (EA) among patients with major depressive disorder compared to ACT only and a control group (treatment-as-usual) across three timelines, such as pre-intervention, immediately post-intervention (8 weeks) and 24 weeks post-intervention.
3. To evaluate the efficacy of exergames-acceptance and commitment therapy (e-ACT) training program on reducing severity of anxiety symptoms among patients with major depressive disorder compared to ACT only and a control group (treatment-as-usual) across three timelines, such as pre-intervention, immediately post-intervention (8 weeks) and 24 weeks post-intervention.
4. To assess the differences in biological markers such as BDNF, CRP, and VEGF among patients on exergames-acceptance and commitment therapy (e-ACT) training program, ACT only and control group (treatment-as-usual) via blood biochemical analyses, at 3 timelines (pre-intervention, immediately post-intervention [8 weeks] and 24 weeks post-intervention).

Research design:

This randomized controlled trial (RCT) is multicentre, three-armed, parallel-group, double-blind RCT.

Study area:

This RCT is expected to run for a duration of 3 years to be conducted in Psychiatric Outpatient clinic in Advanced Medical and Dental Institute, Universiti Sains Malaysia (AMDI, USM) and Psychiatric Outpatient clinic and Inpatient wards in Department of Psychiatry, Hospital Universiti Sains Malaysia (HUSM). AMDI, USM is a tertiary referral centre in which its psychiatry out-patient clinic has approximately 200 registered psychiatric patients in the northern region of Peninsular Malaysia. While HUSM is a tertiary referral centre in which the Department of Psychiatry has approximately 500 to 700 registered psychiatric patients located in the northeast region of Peninsular Malaysia.

Study population:

This study's participants will be recruited from the source population. This population includes all patients diagnosed with major depressive disorder and registered in AMDI, USM and Department of Psychiatry, HUSM.

Sample size estimation:

The sample size is determined based on G-Power 3.1.9.2 for repeated measures, between-within interaction ANOVA. Based on the previous study, the sample size was calculated based on a multicentre, three-group parallel, RCT which compared efficacy of physical exercise, cognitive behavioral therapy and treatment-as-usual control group conducted by Hallgren et al. (2018), with small effect size (0.13), an alpha error of 0.05, two-tailed. The results indicated that the total sample of 90 for three equal-sized groups is needed to achieve a power of 0.95. In anticipation of a drop-out rate of 30%, the estimation for sample size is 117 respondents and hence, we round up to 120 subjects for the total respondents needed. Therefore, 40 respondents for each group.

Sampling method and subject recruitment:

The sampling method use in this study for recruitment of participants is by consecutive sampling.

Recruitment of subjects:

This study's participants will be recruited from the source population. This population includes all patients diagnosed with major depressive disorder and registered in AMDI, USM and Department of Psychiatry, HUSM. These patients will be approached by the research team and explained on the study objectives and procedures. Those who are interested to participate in the study will be screened for inclusion and exclusion criteria.

All eligible patients (those with all inclusion criteria without any exclusion criteria) will be invited to participate in this study. The study's purposes and procedures will be thoroughly explained (verbal explanation by the research assistant and a copy of the participant information will also be distributed) to prospective participants before they are invited to participate in this study, their anonymity will be assured, and they will be informed of their right to withdraw from the study at any time and the data collected will be discarded. Eligible patients will be given 48 hours to decide on their participation in the study. Then, participants will sign written informed consent to participate in the study before they enrol in the study.

Intervention:

An eight-week psychosocial intervention will be administered to participants in each intervention group (e-ACT and ACT) while participants in the control group will receive treatment-as-usual. The study's outcomes will be assessed at three times: pre-intervention (t0), immediately after the eight-week intervention (t1), and 24 weeks after the intervention (t2). Both the e-ACT and ACT interventions will comprise eight sessions delivered at a rate of one session per week.

1. exergames-acceptance and commitment therapy (e-ACT) training program: In the e-ACT training program, participants will perform a 30-minute per session Nintendo-program on TV for three days per week and a 50-minute ACT session per week for 8 weeks which will take place in the psychology labs of AMDI, USM. The ACT session will be held after 30 minutes break following the completion of the final exergame session of the week. Hence, the total duration of each weekly e-ACT training session will be approximately 2 hours. In addition, each weekly e-ACT training session will be held at the same time (± 2 hours) and at the same venue.
2. Acceptance and commitment therapy (ACT):

   As for the ACT intervention, each ACT session will run for 50 minutes, one session per week for 8 weeks. Each weekly ACT session will be held at the same time (± 2 hours) and at the same venue (in the psychology lab).
3. Treatment-as-usual control (TAU) group:

The participants in the control group will receive treatment-as-usual in which non-specific ingredients of the psychotherapeutic approach will be administered, such as psychological understanding to the management of an individual patient, identifying current problems, providing opportunities for disclosure, reassurance, and deep breathing exercise. They will be given equal amount of time and attention from the professional figure compared to the intervention groups, whereby they will also attach to an 8-session program (with one session per week for 8 weeks). Each weekly TAU session will be held at the same time (± 2 hours) and at the same venue (in the psychology lab).

Blinding:

Participants will be kept unaware of the study's randomization into the designated groups, conducted by a research assistant who is not otherwise involved in the study and concealed in an opaque, sequentially numbered envelope. Therefore, participants will not know which group they are allocated to. In addition, the intervention groups (e-ACT or ACT) as well as the treatment-as-usual control group will receive an 8-session program (with one session per week for 8 weeks) and participants in the treatment-as-usual group will also receive equal amount of attention and time from the professional figure who administer the program.

The researchers will also be "blinded" for the study since the participants' randomized assignment into the designated groups will be conducted by a research assistant who is not otherwise involved in the study or data analysis. This project's data collection will also be conducted by that research assistant who is not otherwise involved in the study or data analysis and who is unaware of the study's hypotheses. Moreover, the project's data analysis will be conducted by statisticians who are not otherwise involved in the study. A statistical analysis plan is established prior to the final unblinded of the data lock.

Data collection:

Data collection will be conducted every weekday during working hours, and flyers announcing the study and the benefits of participating in this study will be disseminated to all patients at the study's focal institutions in order to ensure adequate subject enrolment to achieve the calculated sample size. This clinical trial protocol was written according to the "Standard Protocol Items: Recommendations for Intervention Trials 2013." Before the interventions began (t0), the participants will be administered the socio-demographic and clinical characteristics questionnaire, HAMD, MADRS, HAMA, WHOQOL-BREF and AAQ-II. Blood sample will also be collected from all participants to evaluate for the serum level of BDNF, VEGF, and CRP (biomarkers for depression). Then, immediately after the end of the interventions at 8 weeks (t1), assessments with HAMD, MADRS, HAMA, WHOQOL-BREF and AAQ-II is repeated for all participants and blood sample collected for biomarker analysis. Finally, 24 weeks after the completion of the interventions (t2), the questionnaire assessment is repeated for all participants and blood sample collected for biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with major depressive disorder (confirmed by Diagnostic and Statistical Manual for Mental Disorder 5th Edition or DSM V).
2. Those with score of more than 8 based on Hamilton Depression Rating Scale (HAMD).
3. Age 18 to 60 years old
4. Those on a stable medication regimen for at least the past 8 weeks and willing to maintain current treatments throughout the study

Exclusion Criteria:

1. Pregnant women
2. Those who have current and lifetime history of engaging in any psychotherapy
3. Those who consumed alcohol and illicit drugs (Heavy or mild)
4. Those who has current and lifetime history of other psychiatric illnesses, such as other depressive disorders (persistent depressive disorder, premenstrual dysphoric disorder), psychotic disorders (schizophrenia, schizophreniform disorder, schizoaffective disorders, brief psychotic disorder, and delusional disorder), bipolar mood disorder, obsessive compulsive disorder, posttraumatic stress disorder, and attention deficit hyperactive disorder, and autism spectrum disorder
5. Those who are on medications that can induce psychiatric symptoms, such as cardiovascular agents (clonidine, guanethidine, methyldopa, reserpine, beta blockers), dermatologic agents (isotretinoin), anticonvulsants (levetiracetam), antimigraine medications (triptans), hormonal agents (corticosteroids, oral contraceptives, gonadotropin-releasing hormone agonists, tamoxifen), varenicline, immunological agents (interferons), and levodopa
6. Patient who has suicidal tendency

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Rating Scale for Depression score across time points | At three time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after baseline (immediately after completion of intervention), and t2 = 24 weeks after completion of intervention
  The HAMD measures depression in individuals before, during and after treatment. The HAMD is an observer administered instrument. The scale contains 21 items, but is scored based on the first 17 items, which are measured either on 5-point or 3-point scales. Scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression with a maximum score being 52. Studies on the psychometric properties of the HAMD indicated that its has adequate internal consistency where in most studies, its Cronbach's α was > 0.7. It also exhibited good convergent and discriminant validity.

SECONDARY OUTCOMES:
Change in Acceptance and Action Questionnaire score across time points | At three time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after baseline (immediately after completion of intervention), and t2 = 24 weeks after completion of intervention
  The Malay version of the "Acceptance and Action Questionnaire" (AAQ-II) will be used to measure degrees of experiential avoidance or psychological inflexibility among participants. The AAQ-II is the questionnaire's second version, revised from the original version, and it is shorter (seven items) while offering better psychometric consistency. Participants' AAQ-II scores will be calculated by summing up the questionnaire's seven items. Total score could range from 7 to 49. Higher scores indicate higher levels of psychological inflexibility. Validation of the Malay version of the AAQ-II has indicated that the tool has excellent internal consistency with a Cronbach's alpha of 0.91, and it has been found to be a unidimensional scale that measures psychological inflexibility/EA.
Change in World Health Organization Quality of Life Questionnaire-BREF score across time points | At three time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after baseline (immediately after completion of intervention), and t2 = 24 weeks after completion of intervention
  WHOQOL-BREF is a self-administered questionnaire and was used in this study to assess the quality of life of the kratom users. It comprised of 26 items in which items 1 and 2 are general questions on quality of life while the rest of the items are grouped into 4 domains. Each item is scored in a Likert scale ranged from 1-5. WHOQOL-BREF has good psychometric properties and found to be a valid and reliable alternative to WHOQOL-100 for measuring quality of life. The higher the score, the better is the degree of quality of life. The Malay version of the WHOQOL-BREF also demonstrated excellent psychometric properties with internal consistency (Cronbach's α) of 0.89. Each domain is scored from a scale of 0 to 100.
Change in Hamilton Anxiety Scale score across time points | At three time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after baseline (immediately after completion of intervention), and t2 = 24 weeks after completion of intervention
  The HAMA measures anxiety in individuals before, during and after treatment. The HAMA is an observer administered instrument. The tool consists of 14 items, each categorized by a series of symptoms, and measures mental agitation and psychological distress, as well as anxiety-related physical complaints. The responses on the scale were measured on a 5-point Likert scale: 0 (symptoms not present), 1 (mild symptoms), 2 (moderate symptoms), 3 (severe symptoms) and 4 (very severe symptoms). The total score was calculated by summation of the 14 items. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. HAMA exhibited good psychometric properties and widely used for assessment of severity of anxiety symptoms in clinical and research settings.

OTHER OUTCOMES:
Change in serum BDNF (in pg/mL) across time points | At three time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after baseline (immediately after completion of intervention), and t2 = 24 weeks after completion of intervention
  Serum samples will be analyzed for the concentration of protein by commercial enzyme-linked immunoabsorbent assay (ELISA) kit following manufacturer's instructions. Samples may need to be diluted with appropriate amounts of buffer provided in the kit to give constant dilutions prior to analyses. A standard curve will be constructed, and the concentration of samples will be read against the standard curve and expressed as concentration per unit of the samples. The modulation of these immunological parameters will also be determined using gene expression analyses using via real-time PCR.
Change in serum VEGF (in pg/mL) across time points | At three time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after baseline (immediately after completion of intervention), and t2 = 24 weeks after completion of intervention
  Serum samples will be analyzed for the concentration of protein by commercial enzyme-linked immunoabsorbent assay (ELISA) kit following manufacturer's instructions. Samples may need to be diluted with appropriate amounts of buffer provided in the kit to give constant dilutions prior to analyses. A standard curve will be constructed, and the concentration of samples will be read against the standard curve and expressed as concentration per unit of the samples. The modulation of these immunological parameters will also be determined using gene expression analyses using via real-time PCR.
Change in serum C-reactive protein (in mg/L) across time points | At three time points of assessment: t0 (baseline) = before starting intervention, t1 = 8 weeks after baseline (immediately after completion of intervention), and t2 = 24 weeks after completion of intervention
  Serum samples will be analyzed for the concentration of protein by commercial enzyme-linked immunoabsorbent assay (ELISA) kit following manufacturer's instructions. Samples may need to be diluted with appropriate amounts of buffer provided in the kit to give constant dilutions prior to analyses. A standard curve will be constructed, and the concentration of samples will be read against the standard curve and expressed as concentration per unit of the samples. The modulation of these immunological parameters will also be determined using gene expression analyses using via real-time PCR.

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual data will be made available after publication of the study's findings (data such as socio-demographic and clinical characteristics, HAM-D, HAM-A, AAQ-II, WHOQOL-BREF scores, and biological markers serum level (BDNF, VEGF and CRP). The data will be uploaded in Figshare data repository after completion of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Zhang B, Deng H, Ren J, Legrand FD, Ahmad Yusof H, Zhang R, Leong Bin Abdullah MFI. Study protocol on the efficacy of exergames-acceptance and commitment therapy program for the treatment of major depressive disorder: comparison with acceptance and commitment therapy alone and treatment-as-usual in a multicentre randomised controlled trial. BMJ Open. 2024 Jun 26;14(6):e080315. doi: 10.1136/bmjopen-2023-080315. PMID 38926142